CLINICAL TRIAL: NCT05787301
Title: Study of Epidemiologic Investigation and Mechanism of Brain Network of Otologic and Cognitive Function With Post-COVID-19
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-151-01
Record Dates: First submitted 2023-03-21; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Cognitive Decline; Otological Disease
Keywords: COVID-19; Epidemiologic Investigation; Brain network; Otological Symptoms; Cognitive Function
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction; Ear Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with hearing loss after infection: Patients with hearing loss after infection
- Patients with hearing loss before infection: Patients with hearing loss before infection
- Healthy control: Healthy subjects who have never been infected with COVID-19 or diagnosed with hearing loss.

SUMMARY:
The purpose of this study was to analysis the incidence of ear symptoms, cognitive function decline and emotional disorders in Chinese people who were infected with COVID-19, exploring the impact of COVID-19 on the auditory system, cognitive function and emotional function, and analyzing the changes in functional connectivity of brain network after COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cases of COVID-19 that test positive for nucleic acid or antigen
* After infection with COVID-19, the patient has experienced hearing loss, tinnitus, ear tightness, ear pain, vertigo and other ear symptoms, memory loss, depression and so on

Exclusion Criteria:

* Diagnosed cognitive disability
* Patients with confirmed Meniere's disease, auditory neuropathy, and heavy noise exposure
* Those with incomplete basic information or for other reasons are unable to complete questionnaires and other listening and cognitive assessments

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 748 patients with novel coronavirus were surveyed from December 2022 to February 2023.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
The correlation between the peak of COVID-19 transmission and the popularity of related online terms | through study completion, an average of 3 months
  The correlation between the peak of COVID-19 transmission and the popularity of related online terms
Symptom incidence | through study completion, an average of 3 months
  According to the questionnaire survey of 748 patients, the incidence of hearing loss, tinnitus, ear tightness, earache, vertigo or other cognitive and emotional problems after COVID-19 was analyzed.
Pure tone average | through study completion, an average of 3 months
  According to the WHO grading standard of hearing loss in 1980, the average pure tone threshold (PTA) of 0.5k, 1k, 2k and 4kHz in better ears was defined as normal hearing, 26-40 dB HL(hearing level) was defined as mild hearing loss, and 41-55 dB HL was defined as moderate hearing loss. 56-70 dB HL was moderate to severe hearing loss, 71-90 dB HL was severe hearing loss, and ≥91 dB HL was extremely severe hearing loss.
Mini-Mental State Examination score and grade | through study completion, an average of 3 months
  There are 30 points in the Mini-Mental State Examination (MMSE) scale. The score of 27-30 is normal, and 21-26 is mild dementia. 10-20 is moderate dementia; On a scale of 0 to 9, dementia is severe
Montreal Cognitive Assessment score and grade | through study completion, an average of 3 months
  The total score of the Montreal Cognitive Assessment (MoCA) scale is 30 points, generally ≥26 points normal, 18-26 points mild cognitive impairment, 10-17 points moderate cognitive impairment, and < 10 points severe cognitive impairment.
Pittsburgh Sleep Quality Interview score and grade | through study completion, an average of 3 months
  Pittsburgh Sleep Quality Index (PSQI) Scale total scores 21 points. A score of 0-5 indicates good sleep quality; A score of 6-10 indicates good sleep quality; 11-15 points, indicating average sleep quality; A score of 16 to 21 indicates poor sleep quality
Hamilton depression score and grade | through study completion, an average of 3 months
  For the 24th version of Hamilton depression Scale (HAMD), the total score > 35 May indicate severe depression; 21-35, may be mild to moderate depression; 9-20, suspected depression; < 8 indicates normal.
Resting state of Electroencephalogram data | through study completion, an average of 3 months
  Electroencephalogram (EEG) data of the study were preprocessed and trends in functional brain network connectivity were analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China